CLINICAL TRIAL: NCT01246388
Title: Evaluation of Fibrosis and Steatosis in Patients With Chronic Hepatopathy: Non-invasive Imaging and Serum Markers vs. Liver Biopsy
Brief Title: Non-Invasive Evaluation of Fibrosis and Steatosis in Chronic Hepatopathy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tischendorf, Jens, M.D. (Individual)
Responsible Party: Sponsor
Other Study IDs: LU-TI-01
Record Dates: First submitted 2010-10-31; First posted 2010-11-23 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2012-03

CONDITIONS: Chronic Liver Disease; Steatohepatitis; Fibrosis
Keywords: Fibrosis; Steatosis; Liver biopsy; Elastography; MRI
MeSH Terms: conditions — Fatty Liver; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Liver Disease

SUMMARY:
The purpose of this study is to evaluate non-invasive parameters for staging and grading of chronic hepatopathy in comparison to liver biopsy.

DETAILED DESCRIPTION:
For diagnosis, staging and grading of chronic liver disease, liver biopsy is the gold standard to date. Unfortunately, being an invasive diagnostic method, liver biopsy has a significant morbidity. Furthermore, due to the small sample size, sampling error (over- or underestimating severity of liver disease) is a serious problem in diagnostic of chronic liver disease.

The objective of this study is to evaluate non-invasive diagnostic methods (MRI, elastography, ultrasound and serum parameters) in comparison to the gold standard to establish criteria for diagnostic in liver disease and reduce the necessary amount of liver biopsies in the future and allow regular follow up.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatopathy and necessity of liver biopsy

Exclusion Criteria:

* metal implants preventing MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: in- and outclinic patients of the RTWH University Hospital (Department of Medicine III) with chronic hepatopathy and the necessity of undergoing liver biopsy for diagnostic work up
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-05; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Quality of staging fibrosis (METAVIR scoring system) with a combination of MRT and blood serum markers compared to liver biopsy (gold standard) | singular evaluation at the time of liver biopsy (completion of measurements within 2 days before or after liver biopsy)
  Receiver operating characteristic analysis is performed (Area-under-the-ROC-curve) to evaluate non-invasive fibrosis assessment in comparison to the liver biopsy with SPSS-Software, p < 0,05 is regarded as statistically significant. METAVIR is a 5-point scale used in staging fibrosis (0 = no fibrosis, 4 = high grade fibrosis, cirrhosis).

SECONDARY OUTCOMES:
Quality of staging steatosis (four-graded scale, percentage) with a combination of MRT and blood serum markers compared to liver biopsy (gold standard) | singular evaluation at the time of liver biopsy (completion of measurements within 2 days before or after liver biopsy)
  Receiver operating characteristic analysis is performed (Area-under-the-ROC-curve) to evaluate non-invasive steatosis assessment (MR-spectroscopy, ultrasound)in comparison to the liver biopsy with SPSS-Software, p < 0,05 is regarded as statistically significant. The degree of steatosis in liver biopsies and ultrasound is assessed by a morphological semiquantitative approach: 0: none, 1: slight, 2: moderate and 3: severe.

CONTACTS AND LOCATIONS:
Overall Officials: Holger H Lutz, M.D., Principal Investigator — Department of Medicine III, University Hospital RTWH University of Aachen
Locations (1):
- Department of Medicine III, University Hospital Aachen (RWTH), Aachen, Germany

REFERENCES:
- [Background] Castera L. Transient elastography and other noninvasive tests to assess hepatic fibrosis in patients with viral hepatitis. J Viral Hepat. 2009 May;16(5):300-14. doi: 10.1111/j.1365-2893.2009.01087.x. Epub 2009 Feb 25. PMID 19254351
- [Background] Bonekamp S, Kamel I, Solga S, Clark J. Can imaging modalities diagnose and stage hepatic fibrosis and cirrhosis accurately? J Hepatol. 2009 Jan;50(1):17-35. doi: 10.1016/j.jhep.2008.10.016. Epub 2008 Nov 8. PMID 19022517
- [Background] Faria SC, Ganesan K, Mwangi I, Shiehmorteza M, Viamonte B, Mazhar S, Peterson M, Kono Y, Santillan C, Casola G, Sirlin CB. MR imaging of liver fibrosis: current state of the art. Radiographics. 2009 Oct;29(6):1615-35. doi: 10.1148/rg.296095512. PMID 19959511